CLINICAL TRIAL: NCT03219866
Title: Preliminary Study for Comparison of Triple Therapy Nebulizer Versus Dry Powdered Inhaler for Care Transitions in COPD
Brief Title: Nebulizer Versus Dry Powdered Inhalers for Chronic Obstructive Pulmonary Disease (COPD)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lower enrollment than Sponsor expected - Sponsor stopped study
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00042362
Record Dates: First submitted 2017-07-12; First posted 2017-07-18 (Actual); Results first posted 2021-06-10 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2020-09

CONDITIONS: COPD; COPD Exacerbation
Keywords: Nebulizer; Inhaler
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Nebulizers and Vaporizers; Dry Powder Inhalers; Formoterol Fumarate; Budesonide; Ipratropium; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Nebulizers (Experimental): Subjects will receive a long-acting B2-agonist (LABA; Brovana, twice daily), corticosteroid (ICS; Pulmicort, twice daily), and a short-acting anti-cholinergic (SAMA; Atrovent, three times a day).
  Interventions: Device: Nebulizers; Drug: Brovana; Drug: Pulmicort; Drug: Atrovent
- Dry Powder Inhaler (Experimental): Subjects will receive a LABA/ICS (Advair Diskus, twice daily) plus a long-acting anticholinergic (LAMA; Spiriva Handihaler, once daily).
  Interventions: Device: Dry Powder Inhaler; Drug: Advair Diskus; Drug: Spiriva HandiHaler

INTERVENTIONS:
Device: Nebulizers — Patients treated and discharged on nebulized bronchodilators
  Other Names: Nebulizer Arm
  Arms: Nebulizers
Device: Dry Powder Inhaler — Patients treated and discharged on Dry Powder Inhalers
  Other Names: DPI Arm
  Arms: Dry Powder Inhaler
Drug: Brovana — Subjects will receive a long-acting B2-agonist(LABA; Brovana, twice daily)
  Other Names: LABA
  Arms: Nebulizers
Drug: Pulmicort — Subjects will receive a corticosteroid (ICS; Pulmicort, twice daily)
  Other Names: ICS
  Arms: Nebulizers
Drug: Atrovent — Subjects will receive a short-acting anti-cholinergic (SAMA; Atrovent, three times a day)
  Other Names: SAMA
  Arms: Nebulizers
Drug: Advair Diskus — Subjects will receive a LABA/ICS (Advair Diskus, twice daily)
  Other Names: LABA, ICS
  Arms: Dry Powder Inhaler
Drug: Spiriva HandiHaler — Subjects will receive a long-acting anticholinergic (LAMA-Spiriva Handihaler, once daily)
  Other Names: LAMA
  Arms: Dry Powder Inhaler

SUMMARY:
This will be a non-blinded feasibility (pilot) study comparing triple therapy nebulizer vs dry powdered inhalers (DPI) for care transitions in Chronic obstructive pulmonary disease (COPD) exacerbation patients.

We hypothesize that patients treated in hospital and discharged on respiratory medications administered by nebulizers will exhibit better quality of life (QoL), symptom control, and lower COPD and all cause hospital readmission rates compared with patients treated with respiratory medications delivered by DPI.

We aim to demonstrate that:

1. Patients treated and discharged on nebulized bronchodilators will have fewer readmissions to hospital at 30 and 90 days compared to the group utilizing DPI
2. The nebulizer group will demonstrate a longer duration of time until hospital readmission for COPD and all cause readmission compared to the group utilizing DPI
3. The nebulizer group will demonstrate better QoL (measured by the SGRQ - Saint George Respiratory Questionnaire) and symptom control (as measured by the CAT & mMRC) compared to the group utilizing DPI.

DETAILED DESCRIPTION:
Drugs used to treat Chronic obstructive pulmonary disease (COPD) are available primarily in hand held inhaler devices that deliver dry powder (DPI), a soft mist or a metered dose of spray (MDI). The frail, arthritic elderly are often prescribed DPI rather than MDI or soft mist devices, because they require less coordination. DPIs however require the ability to inhale against a resistance with a peak inspiratory force (PIF) more negative than 60 L/min to break the dry powder into respirable particles. Preliminary data suggests that suboptimal PIF's are common during an acute exacerbation of COPD, affecting 48% of hospitalized patients, thus placing them at risk for treatment failure and possibly hospital readmission. Use of nebulizers to administer respiratory medications may avoid the hazards of insufficient dosing that can result from use of DPI however they are cumbersome, expensive and the variety of drugs available in a nebulizer format is limited. We hypothesize that patients treated in hospital and is charged on respiratory medications administered by nebulizers will exhibit better symptom control and lower COPD and all cause hospital readmission rates compared with patients treated with respiratory medications delivered by DPI. We aim to demonstrate that 1) patients treated and discharged on nebulized bronchodilators will have fewer readmissions to hospital at 30 and 90 days compared to the group utilizing DPI 2) that the nebulizer group will demonstrate a longer duration of time till hospital readmission for COPD and all cause readmission compared to the group utilizing DPI and 3) the nebulizer group will demonstrate better symptom control compared to the group utilizing DPI. This nonblinded feasibility (pilot) study will enroll 100 patients hospitalized for an exacerbation of COPD who are > 40 years of age, have a clinical diagnosis of COPD. The study will consist of 3 outpatient visits (Transitional Care Visit [314 days after discharge], Visit #2 [30 +/5 days after discharge], and Visit #3 [90 +/5 days after discharge]). Visit #2 and #3 are for study purposes, the Transitional Care Visit is standard of care. We hypothesize and aim to demonstrate that patients treated in hospital and discharged on respiratory medications administered by nebulizers will exhibit better quality of life (QoL), symptom control and lower COPD and all cause hospital readmission rates compared with patients treated with respiratory medications delivered by DPI.

ELIGIBILITY:
Inclusion Criteria:

* > 40 years of age
* Clinical diagnosis of COPD
* Smoking history > 10 pack years
* Lung Function- FEV1/FVC or FEV1/SVC < 70% on bedside spirometry or previous baseline and FEV1/FVC or FEV1/SVC < 70% on clinic visit < 2 weeks from discontinuation
* Able to give informed consent

Exclusion Criteria:

* Dementia
* Active cancer
* End stage cardiovascular disease
* Inability to attend outpatient visits
* Active Schizophrenia

Pregnancy; subjects will be excluded if female and are not post-menopausal for at least one year. Since there is no possible benefit from participating in this protocol for a pregnant woman, we will exclude pregnant women. If a subject is found to be pregnant during the 90-day study period, they will be excluded from the study and their data not used for study purposes.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill A Ohar, MD, FCCP, Principal Investigator — Professor of Internal Medicine
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). Chronic obstructive pulmonary disease among adults--United States, 2011. MMWR Morb Mortal Wkly Rep. 2012 Nov 23;61(46):938-43. PMID 23169314
- [Background] Pauwels RA, Buist AS, Ma P, Jenkins CR, Hurd SS; GOLD Scientific Committee. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: National Heart, Lung, and Blood Institute and World Health Organization Global Initiative for Chronic Obstructive Lung Disease (GOLD): executive summary. Respir Care. 2001 Aug;46(8):798-825. No abstract available. PMID 11463370
- [Background] Pleasants RA, Ohar JA, Croft JB, Liu Y, Kraft M, Mannino DM, Donohue JF, Herrick HL. Chronic obstructive pulmonary disease and asthma-patient characteristics and health impairment. COPD. 2014 Jun;11(3):256-66. doi: 10.3109/15412555.2013.840571. Epub 2013 Oct 23. PMID 24152212
- [Background] Guarascio AJ, Ray SM, Finch CK, Self TH. The clinical and economic burden of chronic obstructive pulmonary disease in the USA. Clinicoecon Outcomes Res. 2013 Jun 17;5:235-45. doi: 10.2147/CEOR.S34321. Print 2013. PMID 23818799
- [Background] Tashkin DP, Celli B, Senn S, Burkhart D, Kesten S, Menjoge S, Decramer M; UPLIFT Study Investigators. A 4-year trial of tiotropium in chronic obstructive pulmonary disease. N Engl J Med. 2008 Oct 9;359(15):1543-54. doi: 10.1056/NEJMoa0805800. Epub 2008 Oct 5. PMID 18836213
- [Background] Calverley PM, Rabe KF, Goehring UM, Kristiansen S, Fabbri LM, Martinez FJ; M2-124 and M2-125 study groups. Roflumilast in symptomatic chronic obstructive pulmonary disease: two randomised clinical trials. Lancet. 2009 Aug 29;374(9691):685-94. doi: 10.1016/S0140-6736(09)61255-1. PMID 19716960
- [Background] Ferguson GT, Anzueto A, Fei R, Emmett A, Knobil K, Kalberg C. Effect of fluticasone propionate/salmeterol (250/50 microg) or salmeterol (50 microg) on COPD exacerbations. Respir Med. 2008 Aug;102(8):1099-108. doi: 10.1016/j.rmed.2008.04.019. Epub 2008 Jul 9. PMID 18614347
- [Background] Dransfield MT, Bourbeau J, Jones PW, Hanania NA, Mahler DA, Vestbo J, Wachtel A, Martinez FJ, Barnhart F, Sanford L, Lettis S, Crim C, Calverley PM. Once-daily inhaled fluticasone furoate and vilanterol versus vilanterol only for prevention of exacerbations of COPD: two replicate double-blind, parallel-group, randomised controlled trials. Lancet Respir Med. 2013 May;1(3):210-23. doi: 10.1016/S2213-2600(13)70040-7. Epub 2013 Apr 12. PMID 24429127
- [Background] Cazzola M, Page CP, Calzetta L, Matera MG. Pharmacology and therapeutics of bronchodilators. Pharmacol Rev. 2012 Jul;64(3):450-504. doi: 10.1124/pr.111.004580. Epub 2012 May 18. PMID 22611179
- [Background] Cazzola M, Molimard M. The scientific rationale for combining long-acting beta2-agonists and muscarinic antagonists in COPD. Pulm Pharmacol Ther. 2010 Aug;23(4):257-67. doi: 10.1016/j.pupt.2010.03.003. Epub 2010 Apr 8. PMID 20381630
- [Background] Mahler DA, Waterman LA, Gifford AH. Prevalence and COPD phenotype for a suboptimal peak inspiratory flow rate against the simulated resistance of the Diskus(R) dry powder inhaler. J Aerosol Med Pulm Drug Deliv. 2013 Jun;26(3):174-9. doi: 10.1089/jamp.2012.0987. Epub 2012 Oct 1. PMID 23025451
- [Background] Loh CH, Lovings T, Ohar JA . Low Inspiratory Flow Rates Predict COPD and All Cause Readmissions. ATS Abstract;2016;In press

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nebulizers | Dry Powder Inhaler
Started | 21 | 19
Completed | 21 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nebulizers | Dry Powder Inhaler | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 11 | 25
  >=65 years | 7 | 8 | 15
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 61 [57 to 66] | 64 [63 to 73] | 63 [58 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 8 | 23
  Male | 6 | 11 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 5 | 6
  White | 19 | 14 | 33
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 19 | 40
BMI [Mean (Inter-Quartile Range); unit: kg/m2] | 29.9 [22.4 to 33.6] | 25.4 [17.9 to 32.3] | 27.4 [21.4 to 33.2]

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life Measured by St. George's Respiratory Questionnaire (SGRQ)
Description: Scores range from 0 to 100, with higher scores indicating more limitations - Symptoms component (frequency & severity) with a 1, 3 or 12-month recall (best performance with 3- and 12-month recall); Part 2: Activities that cause or are limited by breathlessness; Impact components (social functioning, psychological disturbances resulting from airways disease) refer to current state as the recall
Time Frame: 90 Days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nebulizers | Dry Powder Inhaler
Number analyzed (Participants) | 21 | 19
score on a scale | 49.3 (25.2) | 43.7 (19.8)

2. Secondary Outcome: Symptom Control Measured by the COPD Assessment Test (CAT)
Description: The COPD Assessment Test (CAT) is a patient-completed instrument that can quantify the impact of COPD on the patient's health. The CAT is a validated, short (8-item) and simple patient completed questionnaire. The CAT has a scoring range of 0-40 and a difference or change of 2 or more units over 2 to 3 months in a patient suggests a clinically significant difference or change in health status. A score of >30 indicates that COPD has a very high impact on daily life, a score of >20 indicates a high impact, 10-20 is medium impact, <10 is low impact, and 5 is the upper limit for healthy non-smokers. A higher score would represent a poor outcome for this test.
Time Frame: 90 Days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nebulizers | Dry Powder Inhaler
Number analyzed (Participants) | 21 | 19
score on a scale | 19.2 (9.0) | 16.5 (9.1)

3. Secondary Outcome: Symptom Control Measured by The Modified Medical Research Council Dyspnea Scale (mMRC)
Description: The Modified Medical Research Council Dyspnea Scale, or MMRC, uses a simple grading system to assess a patient's level of dyspnea -- shortness of breath. The scale goes from 0-4 with a 0 = I only get breathless with strenuous exercise, 1 = I get short of breath when hurrying on level ground or walking up a slight hill, 2 = On level ground, I walk slower than people of the same age because of breathlessness or have to stop for breath when walking at my own pace, 3 = I stop for breath after walking about 100 yards or after a few minutes on level ground, and 4 = I am too breathless to leave the house or I am breathless when dressing. 4 would represent the worst outcome.
Time Frame: 90 Days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nebulizers | Dry Powder Inhaler
Number analyzed (Participants) | 21 | 19
score on a scale | 2.1 (1.6) | 1.6 (1.3)

4. Secondary Outcome: COPD and All-Cause Hospital Readmissions After 30 Days
Description: Compare the number of hospital readmissions between the two arms after 30 days of using each device.
Time Frame: 30 Days
Measure: Number; unit: number of readmissions
Arm/Group | Nebulizers | Dry Powder Inhaler
Number analyzed (Participants) | 21 | 19
number of readmissions | 1 | 3

5. Secondary Outcome: COPD and All-Cause Hospital Readmissions After 90 Days
Description: Compare the number of hospital readmissions between the two arms after 90 days of using each device.
Time Frame: 90 Days
Measure: Number; unit: number of readmissions
Arm/Group | Nebulizers | Dry Powder Inhaler
Number analyzed (Participants) | 21 | 19
number of readmissions | 2 | 4

6. Secondary Outcome: Unscheduled Clinic or ER Visits
Description: Compare the number of unscheduled clinic or ER visits between the two arms after 90 days of using each device
Time Frame: 90 Days
Measure: Number; unit: number of visits
Arm/Group | Nebulizers | Dry Powder Inhaler
Number analyzed (Participants) | 21 | 19
number of visits | 4 | 4

7. Secondary Outcome: Change in Pulmonary Inspiratory Force (PIF) From Baseline at 90 Days - R -2 (Low to Medium Resistance Inhalers)
Description: Pulmonary inspiratory force (PIF) from hospital baseline between the two arms for the duration of the 90 day study.
Time Frame: Baseline and 90 days
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Nebulizers | Dry Powder Inhaler
Number analyzed (Participants) | 21 | 19
cmH2O | 73.9 (5.9) | 74.2 (4.2)

8. Secondary Outcome: Number of Deaths
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Nebulizers | Dry Powder Inhaler
Number analyzed (Participants) | 21 | 19
Participants | 1 | 1

9. Secondary Outcome: Change in Pulmonary Inspiratory Force (PIF) From Baseline at 90 Days - R -5 (High Resistance Inhalers)
Description: Pulmonary inspiratory force (PIF) from hospital baseline between the two arms for the duration of the 90 day study.
Time Frame: Baseline and 90 days
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Nebulizers | Dry Powder Inhaler
Number analyzed (Participants) | 21 | 19
cmH2O | 43.7 (2.2) | 46.5 (4.9)

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Nebulizers | Dry Powder Inhaler
All-Cause Mortality (participants affected / at risk) | 1/21 | 1/19
Serious Adverse Events (participants affected / at risk) | 3/21 | 7/19
Other Adverse Events (participants affected / at risk) | 0/21 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nebulizers (N=21) | Dry Powder Inhaler (N=19)
Hospitalizations (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) — Hospitalizations
Re-admissions into Hospital (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) — Re-admissions into Hospital

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/66/NCT03219866/Prot_SAP_001.pdf
  • Informed Consent Form (2020-01-08): https://cdn.clinicaltrials.gov/large-docs/66/NCT03219866/ICF_000.pdf